CLINICAL TRIAL: NCT05276440
Title: Effects of Regional Anesthesia on Postoperative Recovery and Opioid Consumption Following Mastectomy: A Retrospective Study
Brief Title: Effects of Regional Anesthesia Following Mastectomy
Status: Completed | Type: Observational
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Seçil Çetin, Principal Investigator, Koc University Hospital
Other Study IDs: KocUniversity
Record Dates: First submitted 2022-02-19; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General Anesthesia
- Erector Spinae Plane Block
- Rhomboid Block

SUMMARY:
Patients of breast surgery dated between April 2016 and March 2021 will be scanned in three groups; solely induced general anesthesia, general anesthesia induced with Erector Spinae Plane Block, and general anesthesia induced with Rhomboid Block.

The investigators aimed to retrospectively compare the effectiveness of regional anesthesia techniques used in the clinic for postoperative recovery and opioid consumption in patients who underwent breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent breast surgery under general anesthesia with or without one of the blocks; Erector Spinae Plane Block and Rhomboid Block.

Exclusion Criteria:

* Incomplete patient forms.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Breast surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption retrieved from the patient records | up to 24 hours
Length of hospital stay | up to 1 week